CLINICAL TRIAL: NCT01177189
Title: Oxidative Stress Links Aging, Activity and Mobility Limitation
Brief Title: Oxidative Stress Links Aging, Activity, and Mobility Limitation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate effect size.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: E6910-R
Record Dates: First submitted 2010-07-30; First posted 2010-08-06 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2017-09

CONDITIONS: Aging
Keywords: Oxidative Stress; Free radicals; Aging
MeSH Terms: interventions — Thioctic Acid

STUDY DESIGN:
Intervention Model Description: Participants will consume either a daily oral antioxidant cocktail or a placebo. The oral antioxidant cocktail consists of vitamin C, vitamin E, and alpha lipoic acid.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Other): Young healthy men and women aged 18-30
  Interventions: Dietary Supplement: Vitamins C, E, and alpha lipoic acid
- Arm 2 (Other): Older healthy men and women aged >70.
  Interventions: Dietary Supplement: Vitamins C, E, and alpha lipoic acid

INTERVENTIONS:
Dietary Supplement: Vitamins C, E, and alpha lipoic acid — Oral antioxidant cocktail or placebo to be consumed daily

SUMMARY:
The purpose of this study is to understand why and how oxidative stress negatively impacts mobility in the elderly, and to determine whether antioxidant supplements can increase vascular health and mobility.

DETAILED DESCRIPTION:
With the premise that U.S. Veteran demographics reveal an aging population with significant mobility limitation and oxidative stress is tightly linked to both of these characteristics, a series of skeletal muscle/vascular studies are proposed. Specifically, in a series of recent studies the investigators' group has documented positive vascular consequences of antioxidant supplementation during exercise in older subjects that negatively impacted young people. Further provocative findings revealed that following exercise training the older subjects were now also negatively impacted by the antioxidant supplementation. These findings have implications for the understanding of the complex balance between the positive effects of exercise-based rehabilitation, exercise induced oxidative stress, aging, frailty, and subsequent mobility limitation. Therefore four specific aims are proposed that will answer the questions of where (I) oxidative stress is most prevalent in the elderly, why (II) oxidative stress occurs in the elderly, what (III) are the acute consequences of oxidative stress in the elderly, and finally how (IV) can exercise-induced oxidative stress as the result of exercise training in elderly be appropriately managed with exogenous antioxidant therapy to promote compliance and the positive outcome of increased mobility.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged either between 18 - 30 years (young group) and >70 years (old group)
* Free of overt disease. Subjects will be non-obese (BMI < 30) and have plasma glucose concentrations < 7.0 mmol/L under fasting conditions and < 11.1 mmol/L at 120 minutes of an oral glucose tolerance test (OGTT)
* Subjects will be sedentary, defined here as no regular physical activity for at least the prior 2 years
* Candidates must have no orthopedic limitations that would prohibit them from performing cycle or knee-extensor exercise
* All women will be postmenopausal (either natural or surgical) defined as a cessation of menses for at least 2 years, and in women without a uterus, follicle stimulating hormone (FSH) > 40 IU/L

Exclusion Criteria:

* Candidates demonstrating dyslipidemia based on the National Cholesterol Education Program Guidelines of plasma total cholesterol > 240 mg/dl with LDL-cholesterol > 160 mg/dl will be excluded from participation
* Candidates who smoke or are taking medications (blood pressure medications, statins, antioxidants etc.) that could influence the results of the study will not be eligible
* In terms of diet, subjects will be asked to maintain a dietary record for one week prior to the pre-screening and if this reveals a diet that differs substantially from the "typical" average diet in both the young and old, the subject will not be eligible
* Women currently taking hormone replacement therapy (HRT) in the preceding year will be excluded from the proposed studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell S Richardson, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 42 | 45
Completed | 42 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 42 | 45 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 0 | 42
  >=65 years | 0 | 45 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 38
  Male | 21 | 28 | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 45 | 87

OUTCOME MEASURES:

1. Primary Outcome: Vascular Function (i.e. % Flow Mediated Vasodilation)
Description: The effect on flow mediated vasodilation is measured using Doppler ultrasound.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: percentage of vasodilation
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 42 | 45
percentage of vasodilation | 7.4 (0.6) | 5.2 (0.4)

2. Secondary Outcome: Exercise-induced Oxidative Stress (i.e. Free Radical Concentrations and Levels of Lipid Peroxidation)
Description: Free radicals and levels of lipid peroxidation were measured using electron paramagnetic spectroscopy and ELISA assays.
  A minimum value is 0 and a maximum value is 10. A higher value is a worse outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 42 | 45
units on a scale | 1.51 (0.19) | 2.7 (0.13)

3. Secondary Outcome: Vascular Function Following the Antioxidant Intervention
Description: The degree of vasodilation following the antioxidant intervention measured by Doppler ultrasound.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: percentage of vasodilation
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 42 | 45
percentage of vasodilation | 5.8 (0.6) | 8.2 (0.6)

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/45
Other Adverse Events (participants affected / at risk) | 0/42 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT01177189/Prot_SAP_000.pdf